CLINICAL TRIAL: NCT04645329
Title: Should Patients Undergoing Reverse Shoulder Prostheses Due to Arthropathy of the Rotator Cuff be Immobilized? Randomized Prospective Study
Brief Title: Immobilization in Reverse Shoulder Prosthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Carlos Torrens, MD, PhD, Hospital del Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/8752/I
Record Dates: First submitted 2020-11-17; First posted 2020-11-27 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Rotator Cuff Tear Arthropathy
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Intervention Model Description: Randomized prospective study. (computer-generated randomization list and saved in opaque envelopes)
Who Masked: Outcomes Assessor
Masking Description: outcomes assessor will be blinded to the allocation of the patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (no immobilization) (Experimental): patients will be allowed to freely use their arm without any immobilization after surgery
  Interventions: Device: shoulder immovilization sling
- group II (3-week immobilization) (Active Comparator): patients will be kept in an immobilization device for three weeks after surgery
  Interventions: Device: shoulder immovilization sling

INTERVENTIONS:
Device: shoulder immovilization sling — immobilization of the arm after surgery

SUMMARY:
Reverse shoulder prostheses are the treatment of choice in elderly patients with rotator cuff arthropathy. Traditionally these patients have been immobilized for 3 weeks in the immediate postoperative period in order to have good pain control. However, there are no studies that determine the most appropriate period of immobilization. In fact, patients undergoing this type of surgery begin rehabilitation exercises within 24 hours of surgery without experiencing increased pain or requiring specific analgesic treatment. There is a demand in the elderly to limit immobilization time as much as possible, as some live alone and need to be self-sufficient and others have dependents. It would be good to know if it is really necessary to make an immobilization in these patients undergoing this type of surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing primary surgery of inverted prosthesis for rotator cuff arthropathy.
* age between 65-85 a.
* without inflammatory pathologies (rheumatoid arthritis, psoriatic arthritis, ...)
* acceptance to be part of the study.

Exclusion Criteria:

* prosthetic surgery prior to the affected limb.
* other indications of reverse prosthesis other than rotator cuff arthropathies (acute fractures, sequelae fractures, tumor surgery, prosthetic revision surgeries).
* no acceptance to participate in the study.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Pain control (visual analogical scale) | determination of pain the day of the surgery, and then 24hours, 48hours, 7 days, 3-weeks, 3 months, 6 months, 1 year, 2 years postoperatively.
  determination of pain control between groups at different time points with the aid of a visual analogical scale of 10 points, where 0 means no pain and 10 means maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Torrens, MD, PhD, Principal Investigator — Chief Clinic of Parc de Salut Mar
Locations (1):
- Hospital del Mar, Barcelona, Spain